CLINICAL TRIAL: NCT01747551
Title: Randomized, Double-Blind, Placebo Controlled Phase II Study of FOLFOX +/- Ziv-Aflibercept in Patients With Advanced Esophageal and Gastric Cancer
Brief Title: FOLFOX +/- Ziv-Aflibercept for Esophageal and Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-401
Record Dates: First submitted 2012-12-05; First posted 2012-12-11 (Estimated); Results first posted 2018-05-08 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: Advanced
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; aflibercept

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- mFOLFOX6 + Ziv-aflibercept (Active Comparator): Patients received mFOLFOX6 and ziv-aflibercept every 2 weeks. Ziv-aflibercept 4mg/kg was given via intravenous (IV) infusion over 1 hour. Immediately following this was administration of mFOLFOX6: oxaliplatin 85 mg/m2 IV and leucovorin 400 mg/m2 IV were given concurrently over 120 minutes, followed by fluorouracil 400 mg/m2 IV bolus injection and then fluorouracil 2,400 mg/m2 IV infusion over 46 hours. Patients continued on treatment until radiological or clinical progression, unacceptable toxicity, or death.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil; Drug: Ziv-aflibercept
- mFOLFOX6 + Placebo (Active Comparator): Patients received mFOLFOX6 and placebo every 2 weeks. Placebo was given via intravenous (IV) infusion over 1 hour. Immediately following this was administration of mFOLFOX6: oxaliplatin 85 mg/m2 IV and leucovorin 400 mg/m2 IV were given concurrently over 120 minutes, followed by fluorouracil 400 mg/m2 IV bolus injection and then fluorouracil 2,400 mg/m2 IV infusion over 46 hours. Patients continued on treatment until radiological or clinical progression, unacceptable toxicity, or death.
  Interventions: Drug: Oxaliplatin; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: Eloxatin
Drug: Leucovorin
  Other Names: Folinic Acid
Drug: Fluorouracil
  Other Names: 5-FU
Drug: Ziv-aflibercept
  Other Names: ZALTRAP; Eylea
  Arms: mFOLFOX6 + Ziv-aflibercept

SUMMARY:
Anti-angiogenic therapy is a proven therapeutic target in refractory gastric and gastroesophageal junction adenocarcinoma. This trial assessed whether the addition of a high affinity angiogenesis inhibitor, ziv-aflibercept, could improve the efficacy of first-line mFOLFOX6 (oxaliplatin, leucovorin, and bolus plus infusional 5- fluorouracil) chemotherapy in metastatic esophagogastric adenocarcinoma.

In this study (ZAMEGA), patients with treatment-naïve esophagogastric adenocarcinoma were randomly assigned 2:1 in a multicenter, placebo-controlled double-blind trial to receive first-line mFOLFOX6 with or without ziv-aflibercept 4mg/kg every 2 weeks. Randomization was stratified by ECOG performance status (0-1 vs. 2) and primary site of disease (esophagus or GE junction vs stomach).

DETAILED DESCRIPTION:
In patients with esophagogastric cancer, mFOLFOX6 is considered standard of care. Every person has molecules in their bloodstream called vascular endothelial growth factors (VEGFs). These molecules help grow and sustain new blood vessels needed by the human body. Cancer tumors hijack this mechanism because they need new blood vessels and oxygen to grow. Ziv-aflibercept is an antibody, a "targeted therapy" called a "VEGF Trap", that "traps" (binds) these VEGFs and prevents the cancer from using them to grow. Ziv-aflibercept has recently been approved by the FDA for patients with treatment-resistant colorectal cancer. Patients who received standard 5-fluoruracil based chemotherapy pus ziv-aflibercept lived significantly longer than those patients who received standard 5-fluoruracil alone.

The study was designed to have an 80% power, at a 0.20 significance level, to detect a difference in 6-month progression-free survival of 15%, between 65% and 50%. A one-sided log rank test was utilized and all patients treated with at least one dose of mFOLFOX6 and ziv-aflibercept/placebo were included in the statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinoma of esophagus, GE junction or gastric origin
* Disease is not amenable to curative resection and is unresectable, locally advanced or metastatic
* Have not received any prior chemotherapy, investigative or biologic agents for esophagogastric cancer except in the neoadjuvant or adjuvant setting
* Any major surgery must be completed at least 4 weeks prior to study entry, minor procedures must be completed at least 2 weeks prior to study entry
* Vascular access device insertion should be performed at least 1 week prior to study entry. A central line is recommended for all participants
* Willing to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after the last dose of Ziv-aflibercept/placebo

Exclusion Criteria:

* History of hypertension unless adequately controlled
* Evidence of active bleeding from primary tumor at time of study entry
* Pregnant or breastfeeding
* Squamous cell carcinoma histology
* Prior treatment for advanced or metastatic disease
* Palliative radiation to < 25% of bone marrow must have been completed 2 weeks prior to study entry, palliative RT to > 25% must have been completed 4 weeks prior to study entry
* Known allergy to study agents
* Known dihydropyrimidine dehydrogenase deficiency or thymidylate kinase gene polymorphism predisposing participant to 5-FU toxicity
* History of symptomatic congestive heart failure
* Clinically significant peripheral arterial disease
* Grade 2 or higher sensory or motor neuropathy
* Serious unhealed wound, ulcers or bone fractures
* History of HIV positivity or hepatitis B or C
* History of abdominal fistula, wound dehiscence, GI perforation, intra abdominal abscess, uncontrolled GI bleeding or diverticulitis that required hospitalization within 6 months of study entry
* History of arterial thrombotic events
* History of CNS hemorrhage in past 6 months
* Use of warfarin
* History of prior or synchronous malignancy except if treated with curative intent more than 3 years prior to enrollment, or adequately treated non-melanoma skin cancers, cervical carcinoma in situ or prostatic intraepithelial neoplasia without evidence of prostate cancer
* Uncontrolled non-malignant illness
* Uncontrolled psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2017-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from January 2013 through April 2015.
Period: Overall Study
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
Started | 43 | 21
Completed | 0 | 0
Not Completed | 43 | 21
Not completed — Progressive Disease | 24 | 17
Not completed — Death | 3 | 1
Not completed — Adverse Event | 7 | 1
Not completed — Prolonged Treatment Delay | 2 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Physician Decision | 2 | 1
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all randomized patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo | Total
Number analyzed (Participants) | 43 | 21 | 64
Age, Continuous [Median (Full Range); unit: years] | 62 [32 to 83] | 62 [40 to 79] | 62 [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 37 | 18 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 41 | 18 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS)
Description: 6-month PFS is the percent probability of patients remaining alive and progression-free at 6-months from randomization estimated using Kaplan-Meier methods. PFS was measured as the time from randomization to 1st documented disease progression (PD) or death. Patients alive without PD were censored at the earliest of the date of last progression-free disease assessment or start of non-protocol therapy. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Tumor assessments were performed every 8 weeks and evaluated by independent, blinded radiologists. Patient follow-up was 6 months.
Population: The analysis dataset is comprised of all randomized patients.
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
Number analyzed (Participants) | 43 | 21
percent probability | 60.5 [44.3 to 73.3] | 57.1 [33.8 to 74.9]
Statistical Analysis 1: Comparison: mFOLFOX6 + Ziv-aflibercept vs mFOLFOX6 + Placebo; Test type: Superiority; p = 0.72, Log Rank

2. Secondary Outcome: Grade 4 Treatment-Related Toxicity Rate
Description: The percentage of patients who experienced maximum grade 4 treatment-related adverse event based on CTCAEv4 as reported on case report forms.
Time Frame: Adverse events were collected each cycle on treatment. Patients received a median (range) treatment duration (months) of 6.9 (0-23.3) and 6.4 (0-43.9) for mFOLFOX6/ziv-aflibercept and mFOLFOX6/placebo, respectively.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
Number analyzed (Participants) | 43 | 21
percentage of participants | 11.6 [3.9 to 25.1] | 9.5 [1.2 to 30.4]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of patients achieving complete response (CR) or partial response (PR) on treatment based on RECIST 1.1 criteria. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Tumor assessments were performed every 8 weeks and evaluated by independent, blinded radiologists. Patients received a median (range) treatment duration (m) of 6.9 (0-23.3) and 6.4 (0-43.9) for mFOLFOX6/ziv-aflibercept and mFOLFOX6/placebo, respectively.
Population: The analysis dataset is comprised of all patients with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
Number analyzed (Participants) | 36 | 16
percentage of patients | 61.1 [43.5 to 76.9] | 75.0 [47.6 to 97.2]

4. Secondary Outcome: Duration of Objective Response
Description: Duration of response is the time from date of first documented confirmed objective response to date of first documented progressive disease. Per RECIST 1.1 for target lesions: PD is at least a 20% increase in sum LD, taking as reference the smallest sum on study with at least 5 mm absolute increase. For non-target lesions, progression-free means no new lesions or unequivocal progression on existing non-target lesions or not evaluated.
Time Frame: Tumor assessments were performed every 8 weeks and evaluated by independent, blinded radiologists. Patient follow-up (months) median (range) was 14.5 (1.1-49.8) and 18.8 (0.6-49.8) for mFOLFOX6/ziv-aflibercept and mFOLFOX6/placebo, respectively.
Population: The analysis dataset is comprised of patients who achieved objective response except one patient on the mFOLFOX6+Placebo is missing data.
Measure: Mean (Full Range); unit: months
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
Number analyzed (Participants) | 22 | 11
months | 9.0 [1.4 to 22.0] | 8.0 [1.8 to 16.8]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed day 1 of each cycle. Patients received a median (range) treatment duration (months) of 6.9 (0-23.3) and 6.4 (0-43.9) for mFOLFOX6/ziv-aflibercept and mFOLFOX6/placebo, respectively.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. All remaining events regardless of treatment attribution were classified as Other AEs. Per the source vocabulary (CTCAEv4.0) there is a category "Other, specify" for each system organ class. No further data is available to specify classification beyond this general term.
Arm/Group | mFOLFOX6 + Ziv-aflibercept | mFOLFOX6 + Placebo
All-Cause Mortality (participants affected / at risk) | 2/43 | 0/21
Serious Adverse Events (participants affected / at risk) | 34/43 | 9/21
Other Adverse Events (participants affected / at risk) | 43/43 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 + Ziv-aflibercept (N=43) | mFOLFOX6 + Placebo (N=21)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 0
Cardiac disorders -Other (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders -Other (Gastrointestinal disorders) | 2 | 0
Heart failure (Cardiac disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 21 | 1
Hypotension (Vascular disorders) | 0 | 1
Infections and infestations -Other (Infections and infestations) | 0 | 1
Intracranial hemorrhage (Nervous system disorders) | 1 | 0
Investigations -Other (Investigations) | 0 | 1
Malaise (General disorders) | 1 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 3 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 12 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2
Respiratory, thoracic and mediastinal disorders -Other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 4 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 1
Vascular disorders -Other (Vascular disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
White blood cell decreased (Investigations) | 1 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mFOLFOX6 + Ziv-aflibercept (N=43) | mFOLFOX6 + Placebo (N=21)
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 20 | 9
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Alanine aminotransferase increased (Investigations) | 10 | 4
Alkaline phosphatase increased (Investigations) | 21 | 10
Alkalosis (Metabolism and nutrition disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Anal pain (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 32 | 13
Anorexia (Metabolism and nutrition disorders) | 27 | 8
Anxiety (Psychiatric disorders) | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 19 | 10
Atrial fibrillation (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Bloating (Gastrointestinal disorders) | 4 | 1
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 3 | 0
Blood bilirubin increased (Investigations) | 3 | 2
Blurred vision (Eye disorders) | 1 | 2
Bruising (Injury, poisoning and procedural complications) | 2 | 2
Cardiac disorders - Other (Cardiac disorders) | 1 | 0
Chest pain - cardiac (Cardiac disorders) | 2 | 0
Chills (General disorders) | 2 | 1
Cholesterol high (Investigations) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 26 | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 3
Creatinine increased (Investigations) | 4 | 1
Death neonatal (General disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 1
Depression (Psychiatric disorders) | 4 | 1
Diarrhea (Gastrointestinal disorders) | 25 | 9
Dizziness (Nervous system disorders) | 10 | 4
Dry eye (Eye disorders) | 2 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Dysesthesia (Nervous system disorders) | 27 | 12
Dysgeusia (Nervous system disorders) | 11 | 6
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 19 | 9
Dysphasia (Nervous system disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Edema limbs (General disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Eye disorders - Other (Eye disorders) | 1 | 0
Facial pain (General disorders) | 1 | 1
Fatigue (General disorders) | 37 | 19
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1
Fecal incontinence (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 3 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 2
Flushing (Vascular disorders) | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 | 3
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 13 | 10
Gastrointestinal pain (Gastrointestinal disorders) | 9 | 2
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 | 2
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Growth suppression (Musculoskeletal and connective tissue disorders) | 3 | 0
Haptoglobin decreased (Investigations) | 1 | 2
Headache (Nervous system disorders) | 13 | 1
Heart failure (Cardiac disorders) | 1 | 0
Hematoma (Vascular disorders) | 0 | 2
Hemoglobin increased (Investigations) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 4 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 13 | 1
Hot flashes (Vascular disorders) | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 35 | 16
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatremia (Metabolism and nutrition disorders) | 2 | 1
Hypertension (Vascular disorders) | 36 | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 31 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 6 | 3
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 9 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 3
Hyponatremia (Metabolism and nutrition disorders) | 17 | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 0
Hypotension (Vascular disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1
Infusion related reaction (General disorders) | 3 | 0
Injection site reaction (General disorders) | 1 | 0
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 1 | 1
INR increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 11 | 3
Intraoperative hepatobiliary injury (Injury, poisoning and procedural complications) | 0 | 1
Investigations - Other (Investigations) | 7 | 3
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 4 | 2
Lip pain (Gastrointestinal disorders) | 1 | 0
Localized edema (General disorders) | 3 | 3
Lymphocyte count decreased (Investigations) | 1 | 0
Malaise (General disorders) | 9 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4 | 4
Movements involuntary (Nervous system disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 20 | 6
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 4 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 2 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 32 | 15
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Nervous system disorders - Other (Nervous system disorders) | 2 | 2
Neutrophil count decreased (Investigations) | 17 | 7
Non-cardiac chest pain (General disorders) | 4 | 2
Oral dysesthesia (Gastrointestinal disorders) | 8 | 1
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 9 | 0
Pain (General disorders) | 11 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 6 | 2
Paresthesia (Nervous system disorders) | 1 | 2
Paronychia (Infections and infestations) | 1 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 36 | 16
Pharyngeal necrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 2
Platelet count decreased (Investigations) | 23 | 13
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Presyncope (Nervous system disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 8 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal pain (Gastrointestinal disorders) | 2 | 0
Rectal perforation (Gastrointestinal disorders) | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 2 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Nervous system disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 12 | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 | 1
Skin infection (Infections and infestations) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Stomach pain (Gastrointestinal disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 1 | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular disorders - Other (Vascular disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Vomiting (Gastrointestinal disorders) | 10 | 0
Vomiting (Gastrointestinal disorders) | 0 | 5
Watering eyes (Eye disorders) | 2 | 0
Watering eyes (Eye disorders) | 0 | 1
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 11 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
White blood cell decreased (Investigations) | 8 | 3
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No